CLINICAL TRIAL: NCT01507389
Title: A Single-centre, Open-label Trial Investigating the Pharmacokinetics and the Safety Profile After a Single Dose of Liraglutide in Subjects With Hepatic Impairment and in Subjects With Normal Hepatic Function
Brief Title: Safety of Liraglutide in Subjects With Liver Impairment and in Subjects With Normal Liver Function
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NN2211-1328; 2005-003027-38 (EudraCT Number)
Record Dates: First submitted 2012-01-06; First posted 2012-01-10 (Estimated); Last update posted 2014-12-09 (Estimated); Status verified 2014-12

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — Liraglutide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Mild (Experimental)
  Interventions: Drug: liraglutide
- Moderate (Experimental)
  Interventions: Drug: liraglutide
- Severe (Experimental)
  Interventions: Drug: liraglutide
- Normal (Experimental)
  Interventions: Drug: liraglutide

INTERVENTIONS:
Drug: liraglutide — Single dose of 0.75 mg injected subcutaneously (under the skin)

SUMMARY:
This trial is conducted in Europe. The aim of this trial is to investigate liraglutide in subjects with mild, moderate and severe degrees of hepatic impairment compared with subjects with normal hepatic function.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with normal hepatic function and liver parameters within normal range
* Subjects with stable hepatic impairment classified as Child-Pugh grade A, B or C
* Body Mass Index between 18.5-40.0 kg/m^2 (both inclusive)

Exclusion Criteria:

* Known or suspected allergy to trial product or related products
* Liver transplanted subjects
* Cardiac problems
* Uncontrolled treated/untreated hypertension
* Signs of acute liver insufficiency
* Positive HIV (human immunodeficiency virus) 1+2 antibodies
* Cancer or any clinically significant disease or disorder except for conditions associated with the hepatic impairment
* Impaired renal function
* Smoking of more than 10 cigarettes per day, or the equivalent for other tobacco products
* Habitual excessive consumption of methylxanthine-containing beverages and foods (coffee, tea, soft drinks such as cola, chocolate) as judged by the investigator

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2006-03; Primary Completion 2006-06 (Actual); Study Completion 2006-06 (Actual)

PRIMARY OUTCOMES:
Area under the Curve (0-infinity)

SECONDARY OUTCOMES:
Area under the Curve (0-t)
Cmax, maximum concentration
tmax, time to maximum concentration
t½, terminal half-life
Adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Warsaw, Poland

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com